CLINICAL TRIAL: NCT05603247
Title: SWISSHEART: Prediction and Progression of Heart Failure in Switzerland
Brief Title: The SWISSHEART Failure Network (SHFN)
Acronym: Swissheart
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Geneva (Other); University Hospital, Basel, Switzerland (Other); University of Bern (Other); ETH Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: SHFN Swissheart
Record Dates: First submitted 2022-10-20; First posted 2022-11-02 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure Acute; Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute myocardial infarction (AMI) and acute heart failure (AHF): All patients identified with the respective International Statistical Classification of Diseases and Related Health Problems (ICD) 10th revision codes for AMI and/or the phenotype of "AHF" will undergo detailed medical review to verify patients' diagnosis of AMI and/or AHF according to current European Society of Cardiology (ESC) guidelines that are reflected in the subsequent inclusion criteria.

SUMMARY:
A retrospective cohort study will be conducted on patients who were hospitalized at the University Hospital Basel (USB), University Hospital Bern (Inselspital), University Hospital Geneva (HUG) and the University Hospital Zurich (USZ) with the diagnosis of AMI and/or AHF. Baseline data will be collected in the hospital during treatment will be complemented by a short outcome evaluation.

DETAILED DESCRIPTION:
The SWISSHEART Failure (SHF) Registry collects retrospectively Swiss-wide standardized clinical, laboratory, raw data electrocardiograms (ECG) and transthoracic echocardiographies (TTE) of a large number of patients hospitalized for Acute Heart Failure (AHF) or for Acute Myocardial Infarction (AMI), this latter group being at risk of developing heart failure as a consequence of the AMI episode.

Using state-of-the-art statistics and machine learning (ML)-based analyses, This project aims to improve prediction and prevention of heart failure (HF) in AMI patients and understand progression or regression of HF in AHF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients, age > 18 years
2. Hospitalized with a primary diagnosis of AMI

   a) ST-segment elevation Myocardial Infarction (STEMI) and Non-STEMI (NSTEMI) have to fulfil the 4th universal definition of myocardial infarction.
   * Acute myocardial injury with dynamic cardiac troponin (cTn) changes (at least one value above 99th per-centile URL) AND
   * At least ONE of the following:

     * Symptoms of myocardial ischemia
     * New ischemic ECG changes or new pathological Q waves
     * Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality consistent with ischemic etiology
     * Intracoronary thrombus on angiography (or autopsy) AND/OR
3. Hospitalization with a primary diagnosis of AHF based on the following criteria:

   1. Symptoms: progressive dyspnoea, orthopnoea, paroxysmal nocturnal dyspnoea, AND/OR progressive peripheral oedema, weight gain.

      AND at least TWO of the following:
   2. Signs: basal pulmonary rales AND/OR peripheral oedema, jugular vein dilatation OR
   3. N-terminal prohormone of brain natriuretic peptide (NT-proBNP) within 24 hours >450 pg/ml if age <50 years, >900 pg/ml if age 50-75 years, >1800 pg/ml if age >75 years) OR BNP >400 pg/ml. Cut-offs need to be reduced by 50% in case of severe obesity (BMI >35) OR
   4. Treatment of AHF within 24 h using the following drugs i) increased diuretics. iv furosemide or increased po furosemide or torasemide ii) inotropes (dobutamine, dopamine, levosimendan, milrinone) iii) i.v. or s.l. vasodilators (nitroglycerine, isosorbide dinitrate) iv) vasopressors (norepinephrine) OR e) Echocardiographic features (within 72 hours) -- automated TTE downloads left ventricular ejection fraction (LVEF) <40% or estimated pulmonary artery systolic pressure (PASP) >40 mmHg or increased estimated right atrium pressure (RA) pressure above 10 mmHg (VCI size / resp. motion)

For the control cohort, the inclusion criteria are:

1. Female or male patients, age > 18 years
2. ECG and TTE recording performed within 5 days of each other
3. TTE is labelled as "normal".

Exclusion Criteria:

If a subject fulfills the following exclusion criteria, he/she may not be included: Existence of a documented statement of the patient against the use of his/her clinical data for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients identified with the respective ICD-10 codes for AMI and/or the phenotype of "AHF" will undergo detailed medical review to verify patients' diagnosis of AMI and/or AHF according to current ESC guidelines that are reflected in the subsequent inclusion criteria. As there is no specific ICD-10 coding for AHF, inclusion is based on several criteria including signs and symptoms, lab values, typical drugs and echocardiographic criteria within a specific time window.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-03 (Estimated); Study Completion 2023-03-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with major adverse cardiac events (MACE) until March 2023 | up to 3.5 years after last patient inclusion
  MACE is composed of
  * All-cause death
  * Cardiovascular Death
  * Acute myocardial infarction
  * Hospitalization for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Christian M Matter, MD, Principal Investigator — University of Zurich
Locations (4):
- Switzerland (4):
  - University Hospital Basel, Basel
  - University Hospital, Bern, Bern
  - University Hospital, Geneva, Geneva
  - University Hospital, Zurich, Zurich